CLINICAL TRIAL: NCT06403657
Title: DEcentralize Testing, Education, and Linkage to Care by Using Electronic Best Practice Advisory for Hepatitis B (DETECT-B)
Acronym: DETECT-B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam Viral Hepatitis Alliance (Other)
Collaborators: Le Van Thinh Hospital (Other Government); University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Thanh Van Kim, Co-principal investigator, Pham Ngoc Thach University of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DETECT-B protocol
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Viral Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: There are two periods - pre-implementation (used as control) and implementation. The enhanced model will be rolled out in the implementation phase. The change in hepatitis B testing will be evaluated for effectiveness.
  The enhanced model of hepatitis testing and linkage to care includes three implementation interventions: 1) continued medical education (CME) for primary health providers, 2) electronic health records-based best practice alerts (BPA) for chronic hepatitis B testing, 3) point-of-care HBsAg testing (POC). These implementation interventions will be introduced sequentially and cumulatively every four months for 12 months. For example, during the first 4-month period, only CME is implemented. In the next 4 months, BPA will be introduced, coupled with the ongoing CME. In the last 4 months, POC will be introduced, together with the ongoing CME and BPA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of the enhanced model (Experimental): The enhanced model of hepatitis testing and linkage to care includes three implementation interventions: 1) continued medical education (CME) for primary health providers, 2) electronic health records-based best practice alerts (BPA) for chronic hepatitis B testing, 3) point-of-care HBsAg testing (POC). These implementation interventions will be introduced sequentially and cumulatively every four months for 12 months. For example, during the first 4-month period, only CME is implemented. In the next 4 months, BPA will be introduced, coupled with the ongoing CME. In the last 4 months, POC will be introduced, together with the ongoing CME and BPA.
  Since this implementation study is single-sited, the period before the implementation will be used as a control arm.
  Interventions: Other: An enhanced model of hepatitis B testing and linkage to care

INTERVENTIONS:
Other: An enhanced model of hepatitis B testing and linkage to care — Implementing CME sessions (<50 attendees) at Le Van Thinh Hospital will focus on preventive strategies for hepatitis B (HBV). We'll collaborate with IT to integrate a Best Practice Advisory (BPA) system into the hospital's electronic records for hepatitis B testing reminders. The system prompts healthcare workers when a patient lacks HBV screening notes, ensuring timely education and testing. Also, we'll introduce Point-of-Care (POC) HBsAg testing using SD Bioline HBsAg WB® for efficient screening and counseling, with follow-up to ensure care linkage within two weeks.

SUMMARY:
The overarching goal of this implementation study is to determine if an enhanced model of hepatitis B testing and linkage to care could be integrated into a public healthcare facility. To answer this question, the investigators will

1. evaluate the effectiveness of the implementation program (overall impact or individual components) in increasing the use of testing services and linkage to hepatitis B care and treatment,
2. evaluate implementation fidelity, sustainability, and integration of the implementation study and
3. analyze the costs and cost-effectiveness of the implementation study.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) poses a significant public health challenge, particularly in low-income countries like Viet Nam. Despite the development of various diagnostic and treatment tools for hepatitis B, the delivery of these services remains suboptimal.

In response, the investigators seek to assess the feasibility of integrating an enhanced model for hepatitis B testing and linkage to care within a public healthcare facility. The study aims to address this issue through several key objectives:

1. Effectiveness Evaluation: The investigators will evaluate the impact of the implementation program on increasing the utilization of testing services and linkage to hepatitis B care and treatment. This includes assessing the overall impact as well as the effectiveness of individual program components.
2. Implementation Fidelity and Sustainability: The investigators aim to evaluate the fidelity of implementation, examine how well the program is executed, and assess its potential for sustainability and integration into routine healthcare practices.
3. Cost and Cost-Effectiveness Analysis: The investigators will analyze the costs associated with the implementation of the program and its cost-effectiveness in improving hepatitis B testing and linkage to care.

The implementation study is based at Le Van Thinh Hospital in Thu Duc City, Ho Chi Minh City. This study is guided by the EPIS (Explore - Prepare - Implement - Sustain) conceptual framework, which informs our research development, implementation, and evaluation strategies.

A mixed-method quasi-experimental type II hybrid effectiveness-implementation design will be employed. This involves implementing various strategies to enhance hepatitis B testing sequentially over a 12-month period. Strategies include medical education for primary care providers, electronic medical record-based reminders for testing, and point-of-care testing for CHB.

Effectiveness will be assessed using interrupted time series analysis with electronic medical record data. Sustainability will be gauged through interviews or focus group discussions with healthcare providers and patients. Cost evaluation will utilize activity-based costing and cost-effectiveness analysis.

The study aims to generate evidence on the effectiveness and implementation of an enhanced model for hepatitis B screening and care linkage within a primary care setting at a public hospital. The findings are anticipated to be applicable to similar settings in Viet Nam and other lower-middle-income countries globally.

ELIGIBILITY:
Inclusion criteria for patients

* Patients who visit the outpatient clinics at Le Van Thinh Hospital during the study period.
* Consent to use point-of-care HBsAg testing after being fully informed by the health care providers (this only applies during the last 4-month period where POC-HBsAg testing is introduced).

Exclusion criteria for patients: None

Inclusion criteria for healthcare providers and leaders

* Healthcare providers who work in the outpatient department and are involved in the enhanced model during the 12-month implementation period.
* Leaders who are involved in the enhanced model or make decisions or are authorized to to so relating to the enhanced model.
* Consent to join the in-depth interview or focus group after being fully informed by the study investigators.

Exclusion criteria for healthcare providers and leaders: None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in number or proportion HBsAg testing at primary care clinics between pre- and implementation periods, extracted from electronic health records at Le Van Thinh hospital. | Up to 2 years (start one year before the implementation of the enhanced model and end one year after).
  The primary care clinics include general internal medicine clinics and family medicine clinics, located in the outpatient department.
Sustainability of the implementation of the enhanced model, as assessed by EPIS-based semi-structured/structured questionnaires. | At Month 12 of the implementation period
  This is a qualitative outcome. The information will be collected through focus group discussions or in-depth interviews on healthcare staff. The EPIS (Exploration-Preparation-Implementation-Sustainment) is a conceptual framework used to guide the questionnaire and the discussions/interviews
Activity-based costs | At Month 12 of the implementation period
  The scope of the costing was limited to program implementation costs.

SECONDARY OUTCOMES:
Change in linkage to hepatitis B care between pre- and implementation periods, extracted from electronic health records at Le Van Thinh hospital. | Up to 2 years (start one year before the implementation of the enhanced model and end one year after).

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Kim, MD, Principal Investigator — Pham Ngoc Thach University of Medicine

IPD SHARING:
Plan to Share IPD: No